CLINICAL TRIAL: NCT01531699
Title: An Open-label Study to Assess the Antimicrobial Efficacy of ALT005 Ophthalmic Prep Solution (ALT005) Compared to Control (Sterile Saline) Following Dermal Administration in Healthy Volunteers
Brief Title: Antimicrobial Efficacy of ALT005 Ophthalmic Prep Solution in Healthy Volunteers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Altacor Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ALT005/09CL/11/06
Record Dates: First submitted 2012-02-09; First posted 2012-02-13 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Infection Secondary to Surgical Procedure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ALT005 Ophthalmic Prep Solution (Experimental)
  Interventions: Drug: ALT005 Ophthalmic Prep Solution
- saline control (Placebo Comparator)
  Interventions: Other: saline control
- Comparator Product (Experimental): Betadine ophthalmic prep solution
  Interventions: Drug: Betadine ophthalmic prep solution

INTERVENTIONS:
Drug: ALT005 Ophthalmic Prep Solution — single application for up to 6 hours
  Arms: ALT005 Ophthalmic Prep Solution
Other: saline control — single application for up to 6 hours
  Arms: saline control
Drug: Betadine ophthalmic prep solution — single application for up to 6 hours
  Arms: Comparator Product

SUMMARY:
This is an open-label, randomized, single-dose, placebo-controlled efficacy study to assess the antimicrobial efficacy of ALT005 ophthalmic prep solution following dermal administration in healthy volunteers. Efficacy will be assessed by comparing the reduction in microbial load for up to 6 hours to that of saline control.

DETAILED DESCRIPTION:
A total of 45 subjects who meet the criteria for inclusion will receive either ALT005 or control solution (sterile 0.9% saline) on one occasion to sites on the forehead and the cheeks. Subjects will be randomized in a ratio of 2:1 active:control. Subjects will be dosed in groups.

The study will run at one study center in the US. Subjects will be housed in the clinical research facility from the morning of Day -4 until the evening of Day 1. The total duration of participation for each subject dosed is approximately 21 days (from Day -19 study orientation through the follow-up call on Day 2, excluding the initial screening period).

In this study, the efficacy of ALT005 will be assessed in healthy volunteers who, after refraining voluntarily from using topical and oral antimicrobials for at least 2 weeks (14 days), exhibit acceptably high normal flora counts on the designated skin testing sites.

An additional cohort was added (3 ALT005, 6 Comparator Product) to make a non-statistical comparison of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy with no clinically significant findings in the screening results
* Non-tobacco/nicotine-containing product users
* Acceptably high normal (>3 log10) flora counts from the designated skin sites on Day -4.
* Voluntarily consent to participate in the study.
* Females reporting spontaneous postmenopausal status
* WOCBP must either be sexually inactive (abstinent) for 14 days prior to screening and remain so through 30 days following administration (topical dosing) of the study drug or have been using acceptable methods of birth control for the times specified
* WOCBP who have undergone sterilization procedures 6 months prior to Day 1

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic (including sensitive skin on the face), neurological, or psychiatric disease, or any other clinically significant disease not deemed acceptable by the PI.
* Evidence of compromise to skin integrity of forehead or cheek caused by acute rash, exacerbation of dermatitis, exacerbation of acne, or any other acute condition deemed clinically significant by the PI.
* Tattoo, scar, keloid, or other chronic skin condition located on forehead or cheek
* Facial hair growth that would interfere with sample collection procedures.
* Positive urine drug/alcohol or cotinine testing
* Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV).
* History or presence of alcoholism or drug abuse within the 2 years prior to Day 1.
* Hypersensitivity or idiosyncratic reaction to any ingredients in ALT005.
* Use of any prescription medication started within 90 days prior to Day 1
* Use of any over-the-counter (OTC) medication, including herbal products, within the 14 days prior to the Day 1
* Blood donation or significant blood loss within 56 days prior to Day 1
* Plasma donation within 7 days prior to Day 1
* Participation in another clinical trial within 30 days prior to Day 1
* Females who are pregnant or lactating, or have a positive pregnancy test at screening or check-in
* Failure to comply with the pre-treatment restrictions related to showering/washing and contact with antimicrobial substances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
3 log10 reduction in microbial load | 10 minutes post dose
  3 log10 reduction in microbial load at 10 minutes following application to the forehead or cheek compared to Day 1 baseline.

SECONDARY OUTCOMES:
3 log10 reduction in microbial load | 45 minutes post dose
  3 log10 reduction in microbial load at 45 minutes following application to the forehead or cheek compared to Day 1 baseline.
3 log10 reduction in microbial load | 6 hours post dose
  3 log10 reduction in microbial load at 6 hours following application to the forehead compared to Day 1 baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Connolly, MD, Principal Investigator — Celerion
Locations (1):
- Celerion Inc, Neptune City, New Jersey, United States